CLINICAL TRIAL: NCT01412203
Title: Evaluating the Effectiveness of the Dissemination of Action Schools! BC: A Socio-ecological Intervention to Increase Physical Activity and Healthy Eating in School Children
Brief Title: Evaluating the Effectiveness of the Dissemination of Action Schools! BC
Acronym: AS!BC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Victoria (Other); University of Waterloo (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); Ministry of Education, British Columbia (Other); Ministry of Health, British Columbia (Other Government); Ministry of Tourism, Sport and the Arts, British Columbia (Other); Provincial Health Services Authority British Columbia (Other); JW Sporta (Unknown); 2010 Legacies Now (Other)
Responsible Party: Principal Investigator, Heather McKay, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H05-80505
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Physical Activity; Obesity; Physical Fitness
Keywords: Physical activity; Healthy weight; Healthy eating; Physical fitness; Children; School based; Community based; Obesity; Health promotion; Socio-ecological; Environment based
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Practice (No Intervention): School continues with regular programming
- Action Schools! BC (Experimental): School adopts the AS!BC model
  Interventions: Behavioral: Action Schools! BC

INTERVENTIONS:
Behavioral: Action Schools! BC — AS! BC applies a socioecological, whole school approach to promote healthy living within the elementary school context. Schools are provided with the tools and support needed to create customized action plans that promote physical activity (PA) and healthy living across six Action Zones (School Environment, Scheduled Physical Education (PE), Classroom Action, Family and Community, Extra-curricular, School Spirit). Generalist teachers receive training and resources to implement their Action Plan with the ultimate goal of providing students with 150 minutes of PA/week. The model is choice-based; teachers are asked to provide 15 additional minutes of PA/day within the Classroom Action Zone. The activities require minimal equipment and can be performed in the classroom, hallway or on the school playground.
  Arms: Action Schools! BC

SUMMARY:
Childhood obesity is a major public health threat. Physical activity and healthy eating contribute to the maintenance of healthy weights. Individually oriented behaviour change programs may not be able to overcome the influence of what has been called an obesogenic environment. Action Schools! BC (AS! BC) used a socio-ecological approach to enhance opportunities for physical activity and healthy eating in elementary schools and created systemic change at the provincial level. AS! BC helps elementary schools customize action plans, based upon their local context, to contribute to the health and well-being of children and the school community. Pilot research showed that AS! BC was an effective and feasible model. The provincial dissemination of AS! BC has been launched and partners from across many sectors are involved to enhance the sharing of knowledge and increase the implementation of the AS! BC model across British Columbia. The dissemination provides an unprecedented opportunity for evaluating how changing the school environment can promoted healthy weights in children. The dissemination was evaluated using a cluster randomized design; 30 elementary schools (n = 1529 consented children) from four (out of five) provincial health authorities volunteered to participate.

The primary goals of the research are:

1. to determine if the Action Schools! BC (AS! BC) model is an effective approach to positively change school environments and health related behaviours of children from diverse geographical regions and cultural groups, and
2. to determine if the supports provided to schools or the community context influence the uptake and use of the AS! BC model.

This research will contribute to the science of obesity prevention and knowledge use as well as public health practice.

ELIGIBILITY:
Inclusion Criteria:

* Student attends a school that has agreed to participate in the study
* Student's classroom teacher has agreed to participate in the study
* Student is in grade 4 or 5 at start of study
* Student participates in regular physical education classes at school
* Student's parents provide consent

Exclusion Criteria:

* Student does not attend a school that has agreed to participate in the study
* Student's classroom teacher does not agree to participate in the study
* Student is not in grade 4 or 5 at start of study
* Student does not participate in regular physical education classes at school
* Student's parents do not provide consent

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1529 (Actual)
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Physical activity opportunities delivered (minutes/week)
  School level; as measured by Weekly Teacher Logs and Interim Reports
School environment scores
  School level; as measured by a modified School Health Inventory
Height (cm)
  Student level
Weight (kg)
  Student level
Body mass index (kg/m^2)
  Student level
Physical fitness (Fitnessgram (C))
  Student level
Children's leisure time physical activity (PAQ-C)
  Student level
Children's dietary intake
  Student level; 24 hour recall and food frequency survey
Physical activity interventions planned
  School level; as measured by Action Plans

SECONDARY OUTCOMES:
Contextual factors surrounding the use of the intervention
  School level
  * School and community partnership survey
  * Annual focus groups with school planning teams, regional advisory committees, parent advisory committees, the local healthy living alliance
  * Semi-structured telephone interviews with school administrators, AS! BC regional facilitators, public health nursing staff, local nutritionist, municipal recreation staff and representatives of non-government organizations involved in chronic disease prevention locally
  * Review of AS! BC annual reports and action plans
  * Participant observation form to assess development of communities of practice

CONTACTS AND LOCATIONS:
Overall Officials: PJ Naylor, PhD, Principal Investigator — University of Victoria; Heather A McKay, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - University of British Columbia - Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - University of Victoria, Victoria, British Columbia

REFERENCES:
- [Background] Naylor PJ, Macdonald HM, Reed KE, McKay HA. Action Schools! BC: a socioecological approach to modifying chronic disease risk factors in elementary school children. Prev Chronic Dis. 2006 Apr;3(2):A60. Epub 2006 Mar 15. PMID 16539801
- [Background] Naylor PJ, Macdonald HM, Zebedee JA, Reed KE, McKay HA. Lessons learned from Action Schools! BC--an 'active school' model to promote physical activity in elementary schools. J Sci Med Sport. 2006 Oct;9(5):413-23. doi: 10.1016/j.jsams.2006.06.013. Epub 2006 Aug 1. PMID 16884957
- [Derived] Nettlefold L, Naylor PJ, Macdonald HM, McKay HA. Scaling up Action Schools! BC: How Does Voltage Drop at Scale Affect Student Level Outcomes? A Cluster Randomized Controlled Trial. Int J Environ Res Public Health. 2021 May 13;18(10):5182. doi: 10.3390/ijerph18105182. PMID 34068235
- [Derived] McKay HA, Macdonald HM, Nettlefold L, Masse LC, Day M, Naylor PJ. Action Schools! BC implementation: from efficacy to effectiveness to scale-up. Br J Sports Med. 2015 Feb;49(4):210-8. doi: 10.1136/bjsports-2013-093361. Epub 2014 Oct 13. PMID 25312876
- [Derived] Nettlefold L, McKay HA, Naylor PJ, Bredin SS, Warburton DE. The relationship between objectively measured physical activity, sedentary time, and vascular health in children. Am J Hypertens. 2012 Aug;25(8):914-9. doi: 10.1038/ajh.2012.68. PMID 22673018
- See also: Intervention website — http://www.actionschoolsbc.ca/